CLINICAL TRIAL: NCT00711308
Title: Long Term Subcutaneous Tinzaparin Compared With Tinzaparin and Oral Anticoagulants in the Treatment of the Acute Pulmonary Embolism
Brief Title: Tinzaparin in the Treatment of the Acute Pulmonary Embolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Complejo Hospitalario Xeral-Calde (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Pérez de Llano, Luis MD, Pneumology Service, Complejo Hospitalario Xeral-Calde
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EX0401ES; eudract-no. 2004-002019-97
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Acute Pulmonary Embolism
Keywords: pulmonary embolism; low molecular weight heparin; vitamin K antagonist; Longterm
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tinzaparin; Acenocoumarol; acarboxyprothrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tinzaparin (Experimental): tinzaparin (innohep®)subcutaneously in a fixed dose of 175 IU anti-Xa/kg of body weight once daily for 6 months
  Interventions: Drug: tinzaparin
- acenocoumarol (Active Comparator): tinzaparin followed by acenocoumarol for 6 months
  Interventions: Drug: tinzaparin; Drug: acenocoumarol

INTERVENTIONS:
Drug: tinzaparin — tinzaparin (innohep®)subcutaneously in a fixed dose of 175 IU anti-Xa/kg of body weight once daily for 6 months
  Other Names: innohep
Drug: acenocoumarol — acenocoumarol for 6 months
  Other Names: vitamin K antagonist
  Arms: acenocoumarol

SUMMARY:
The purpose of this study is to evaluate the feasibility of the long-term treatment of pulmonary embolism with tinzaparin compared to oral anticoagulants.

DETAILED DESCRIPTION:
The open-label prospective randomized clinical trial compares subcutaneous LMWH (tinzaparin) administered for 6 months versus initial treatment using subcutaneous LMWH followed by oral anticoagulants given for 6 months in patients with acute venous thrombosis.

To evaluate the direct and indirect cost of each treatment regimen in a rural population environment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pulmonary embolism patients confirmed by:

  * High probability ventilation/perfusion lung scan according to the PIOPED criteria
  * Spiral chest computed tomography, or
  * Pulmonary arteriography
* Aged 18 years or above, of either sex
* The patient must provide signed informed consent
* Patients will be agreed for receiving ambulatory anticoagulant treatment

Exclusion Criteria:

* Massive pulmonary embolism
* Allergy to heparin, other components of Tinzaparin or acenocoumarol
* Previous thrombocytopenia induced by heparin
* Thrombocytopenia < 100000/mm3
* History/signs/symptoms of congenital bleeding disorder
* Life expectancy less than 90 days
* Unfractioned heparin anticoagulation for more than 36 hours prior enrollment
* Inability to participate in the home tinzaparin program
* Clinical overt gastrointestinal blood loss due to peptic ulcer, intestinal tumours, oesophagitis or diverticulosis
* Hemoglobin lower than 7 g/dL or Creatinin > 3mg/dL
* Cerebral-vascular accident
* Cerebral, medullary and ophthalmological surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-04; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of the secondary prophylaxis of pulmonary embolism with tinzaparin | 6 months

SECONDARY OUTCOMES:
direct and indirect cost of each treatment regimen | 6 months
Major haemorrhagic events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Luis Pérez de Llano, MD, Study Chair — Complejo Hospitalario Xeral Calde (Lugo); Alejandro Veres Racamonde, MD, Principal Investigator — Complejo Hospitalario Xeral Calde (Lugo); Manuel Núnez Delgado, MD, Principal Investigator — Hospital do Meixoeiro (Vigo); Ana Palacios Bartolomé, MD, Principal Investigator — Hospital Clínico de Santiago; Virginia Leiro Fernández, MD, Principal Investigator — Hospital Xeral (Vigo)
Locations (4):
- Spain (4):
  - Pneumology Service. Hospital Clínico, Santiago de Compostela, A Coruña
  - Pneumology Service, Lugo, Lugo
  - Pneumology Service. Hospital Xeral Cies, Vigo, Pontevedra
  - Pneumology Service. Hospital do Meixoeiro, Vigo, Pontevedra